CLINICAL TRIAL: NCT05149755
Title: Evolut™ EXPAND TAVR II Pivotal Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D00411092
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Moderate Aortic Valve Stenosis
Keywords: aortic; stenosis; moderate; valve; TAVR
MeSH Terms: conditions — Constriction, Pathologic; Lymphoma, Follicular | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Medtronic Evolut PRO+, or Evolut FX,TAVR System, & guideline-directed management & therapy (GDMT) (Experimental): Medtronic Evolut PRO+ TAVR or Evolut FX TAVR Systems, & guideline-directed management & therapy
  Interventions: Device: Medtronic Evolut PRO+ TAVR System, or Evolut FX TAVR System, and guideline-directed management and therapy (GDMT)
- Clinical site determined guideline-directed management and therapy (GDMT) alone (No Intervention): Clinical site determined guideline-directed management and therapy (GDMT) alone

INTERVENTIONS:
Device: Medtronic Evolut PRO+ TAVR System, or Evolut FX TAVR System, and guideline-directed management and therapy (GDMT) — Patients will have a Transcatheter Aortic Valve Replacement (TAVR) with either an Evolut PRO+ TAVR, or Evolut FX TAVR, heart valve, and given clinical site-determined guideline-directed management and therapy (GDMT).
  Arms: Medtronic Evolut PRO+, or Evolut FX,TAVR System, & guideline-directed management & therapy (GDMT)

SUMMARY:
Obtain safety and effectiveness data to support indication expansion for the Medtronic TAVR System to include patients with moderate, AS.

DETAILED DESCRIPTION:
Multi-center, international, prospective, randomized study. Subjects will be randomized to either transcatheter aortic valve replacement (TAVR) with the Evolut PRO+ TAVR System, or Evolut FX System, and guideline-directed management (GDMT) or GDMT alone.

ELIGIBILITY:
Key Inclusion Criteria:

o Moderate AS, defined as follows by transthoracic echo (TTE) as assessed by the ECL:

* AVA >1.0 cm² and <1.5cm²; or
* AVA ≤ 1.0 cm² with AVAI > 0.6cm²/m² if BMI < 30 kg/m²: or
* AVA ≤ 1.0 cm² with AVAI > 0.5cm²/m² if BMI ≥ 30 kg/m²:

and

* Max aortic velocity ≥ 3.0 m/sec. and < 4.0 m/sec. or
* Mean aortic gradient ≥ 20mmHg and < 40.0 mmHg

Any of the following at-risk features:

* Symptoms of AS, defined as:
* NYHA ≥ Class II, or
* Reduced functional capacity, defined as

  * 6MWT < 300 meters, or
  * < 85% of age-sex predicted METs on exercise tolerance testing (ETT)
* Documented heart failure event or hospitalization for heart failure within 1 calendar year prior to consent
* NT-proBNP ≥ 600 pg/ml (or BNP ≥ 80 pg/ml), or
* Persistent AF or Paroxysmal AF episode within 6 months prior to consent, or
* Elevated aortic valve calcium score (>1200 AU for females and > 2000 AU for males) as assessed by the MDCT core lab, or
* Any of the following by the qualifying TTE as assessed by the ECL:

  * Global longitudinal strain ≤16% (absolute value), or
  * E/e' ≥ 14.0 (average of medial and lateral velocities), or
  * Diastolic dysfunction ≥ Grade II, or
  * LVEF < 60%
  * Stroke Volume Index < 35 ml/m²
* Anatomically suitable for transfemoral TAVR using the Medtronic Evolut PRO+ or Evolut FX system
* The subject and the treating physician agree the subject will return for all required follow-up visits

Key Exclusion Criteria:

* Age < 65 years
* LVEF ≤ 20% by 2-D echo
* Class I indication for cardiac surgery
* Contraindication for placement of a bioprosthetic valve
* Documented history of cardiac amyloidosis

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Composite rate of all-cause mortality, all-stroke, life threatening or fatal bleeding, acute kidney injury, hospitalization due to device or procedure-related complication, or valve dysfunction requiring reintervention. | 30 days
  Life threatening or fatal bleeding is defined as BARC Type 3 or 4 and acute kidney injury is defined as VARC-3 Stage IV.
Composite rate of all-cause mortality, heart failure hospitalization or event, or medical instability leading to aortic valve replacement or re-intervention. | 2 years

SECONDARY OUTCOMES:
Proportion of subjects alive and with moderately improved quality of life (≥ 10 points in KCCQ summary score from baseline) | 1 year
Composite of all-cause mortality and heart failure hospitalizations or events. | 2 years
Composite of all-cause mortality, all-stroke, or unplanned CV hospitalizations | 2 years
Heart failure hospitalizations or events. | 2 years
All-cause mortality | 2 years
Unplanned cardiovascular hospitalizations | 2 years
Days alive and free of unplanned cardiovascular hospitalizations | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sorajja, MD, Principal Investigator — Allina Health System; Josep Rodes-Cabau, MD, Principal Investigator — Fondation IUCPQ; Stephan Windecker, Prof., Principal Investigator — Inselspital, Universitätsspital Bern
Locations (93):
- United States (52):
  - University of Alabama at Birmingham (UAB) Hospital, Birmingham, Alabama
  - Abrazo Arizone Heart Hospital, Phoenix, Arizona
  - HonorHealth Scottsdale Shea Medical Center, Scottsdale, Arizona
  - Los Robles Hospital & Medical Center, Thousand Oaks, California
  - University of Colorado Hospital, Aurora, Colorado
  - Saint Vincents Medical Center, Bridgeport, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - University of Florida, Gainesville, Florida
  - Saint Vincent's Medical Center Riverside, Jacksonville, Florida
  - Orlando Health, Orlando, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Tampa General Hospital, Tampa, Florida
  - Jewish Hospital, Louisville, Kentucky
  - Terrebonne General Medical Center, Houma, Louisiana
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan Health System - University Hospital, Ann Arbor, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Catholic Medical Center, Manchester, New Hampshire
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Englewood Hospital & Medical Center, Englewood, New Jersey
  - Northwell Health, Manhasset, New York
  - The Mount Sinai Hospital, New York, New York
  - Mission Hospital, Asheville, North Carolina
  - Wake Forest University Heatlh Sciences, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Kettering Health Main Campus, Kettering, Ohio
  - Oregon Health & Science University Hospital, Portland, Oregon
  - Lehigh Valley Hospital, Inc, Allentown, Pennsylvania
  - UPMC Pinnacle Harrisburg Campus, Harrisburg, Pennsylvania
  - Monument Health Rapid City Hospital, Rapid City, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Medical City Dallas, Dallas, Texas
  - Texas Health Harris Methodist Hospital Fort Worth, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Methodist Hospital San Antonio, San Antonio, Texas
  - Intermountain Cardiovascular and Thoracic Surgery, Salt Lake City, Utah
  - The University of Vermont, Burlington, Vermont
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Providence Sacred Heart Medical Center & Children's Hospital, Spokane, Washington
  - West Virginia University, Morgantown, West Virginia
  - Aurora Saint Lukes Medical Center, Milwaukee, Wisconsin
- Australia (2):
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch
- Austria (2):
  - University Hospital Sankt Poelten, Sankt Pölten
  - Allgemeines Krankenhaus - Universitätskliniken Wien, Vienna
- CHU de Liege- Hopital du Sart Tilman, Liège, Belgium
- Canada (4):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal Heart Hospital, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ), Québec, Quebec
  - Queen Elizabeth II Health Sciences Centre, Halifax
- France (4):
  - CHU de Rennes - Hôpital Pontchaillou, Rennes, Brittany Region
  - CHRU Brest - Hôpital de la Cavale Blanche, Brest
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Européen Georges Pompidou, Paris
- Germany (6):
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen
  - Universitätsklinikum Bonn, Bonn
  - Kath Saint Johannes-Gesellschaft Dortmund gGmbH Saint Johannes-Hospital Dortmund, Dortmund
  - Herzzentrum Leipzig GmbH, Leipzig
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Klinikum der Universität München - Campus Grosshadern, München
- Galway University Hospitals - University Hospital Galway (UHG), Galway, Ireland
- Israel (2):
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center- Beilinson Hospital, Petah Tikva
- Italy (3):
  - Presidio Ospedaliero Gaspare Rodolico, Catania
  - Ospedale San Raffaele - Milano, Milan
  - IRCCS Policlinico San Donato, San Donato Milanese
- Japan (5):
  - Shonan Kamakura General Hospital, Kanagawa, Kamakura
  - Tokai University Hospital, Isehara, Kanagawa
  - Kawasaki Saiwai Hospital, Kawasaki, Kanagawa
  - Osaka Keisatsu Hospital, Osaka
  - Osaka University Hospital, Osaka
- Netherlands (4):
  - Catharina Ziekenhuis, Eindhoven
  - Universitair Medisch Centrum Groningen, Groningen
  - St Antonius Ziekenhuis, Nieuwegein
  - Erasmus MC, Rotterdam
- Spain (4):
  - Hospital Universitari Clínic de Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Clínico Universitario de Valladolid, Valladolid
- Skanes Universitetssjukhus, Lund, Sweden
- Inselspital - Universitätsspital Bern, Bern, Switzerland
- Saint Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No